CLINICAL TRIAL: NCT00451867
Title: A Randomized Multicenter Double-Blind Clinical Trial to Evaluate the Efficacy and Safety of Mycophenolate Mofetil (CellCept) for the Treatment of Refractory Interstitial Cystitis (IC)
Brief Title: A Randomized Multicenter Double-Blind CT to Evaluate the Efficacy and Safety of Mycophenolate Mofetil . . .
Acronym: ICCRN RCT2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The major and primary reason for the study termination is the observed reduced efficacy of CellCept compared to placebo.
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: LeRoy M. Nyberg, PhD., MD, NIDDK
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DK765209-Cellcept (IND)
Record Dates: First submitted 2007-03-23; First posted 2007-03-26 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Interstitial Cystitis; Painful Bladder Syndrome
Keywords: interstitial cystitis research; painful bladder syndrome research; pelvic pain research; interstitial cystitis and autoimmune; interstitial cystitis and cellcept; interstitial cystitis and mycophenolate mofetil; interstitial cystitis and MMF; interstitial cystitis and inflammation; inflammatory diseases and immunosupression
MeSH Terms: conditions — Cystitis, Interstitial; Inflammation | interventions — Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): 2000 mg per day of CellCept (MMF) divided into 2 equal doses.
  Interventions: Drug: Mycophenolate Mofetil; Drug: Mycofenolate Mofetil (MMF)
- B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mycophenolate Mofetil
  Other Names: CellCept
  Arms: A
Drug: Mycofenolate Mofetil (MMF) — 2000 mg per day divided into 2 equal doses.
  Other Names: CellCept
  Arms: A
Drug: Placebo — Placebo
  Arms: B

SUMMARY:
The purpose of this study is to investigate the safety and effectiveness of a medication called CellCept in treating refractory (has not responded to other treatments) interstitial cystitis.

CellCept belongs to a class of medications called immuno-suppressants. Immuno-suppressants work in the body by reducing the immune system's ability to produce certain reactions that can cause inflammation. In some people, the inflammation produced by their immune system can damage healthy tissues and cause symptoms of pain and discomfort. CellCept is approved by the U.S. Food and Drug Administration (FDA) for use in patients who have had an organ transplant. When used in combination with other drugs, CellCept helps to prevent the rejection of the transplanted organ and is used widely in patients who have received kidney, liver and heart transplants. CellCept is also frequently used but not FDA approved for the treatment of severe rheumatoid arthritis which is a disease caused when the body's immune system acts against healthy tissues in the joints.

Due to its special activity, CellCept may be useful in treating certain inflammatory diseases or conditions like interstitial cystitis.

DETAILED DESCRIPTION:
Interstitial Cystitis (IC) is a bladder syndrome characterized as painful, debilitating and chronic, with no universally successful treatment option currently available. Characteristic symptoms include pain with bladder filling, and marked urinary frequency (to relieve pain). The only FDA-approved oral medication for treatment of IC is pentosan polysulfate (Elmiron), recently demonstrated by our collaborative research network to perform with little more efficacy than placebo (ref), and which is expensive and has associated side effects. Current clinical treatment protocols are empiric and usually aimed at relieving pain. There is a pressing need for an effective oral medication for treatment of IC. The presentation of symptoms can be quite variable among patients, suggesting that IC is a multi-factorial syndrome with several proposed etiologies, some of which may be interrelated.

ELIGIBILITY:
Inclusion Criteria:

* Participant at least 18 years of age and received a diagnosis of PBS/IC, confirmed by cystoscopy and hydrodistention in the past with findings of glomerulations and/or ulceration.
* Participant has symptoms of urinary frequency and pain/discomfort (at least 4 on each 0-10 Likert scale) at entry.
* Participant failed at least 24 weeks of active treatment with a minimum of 3 standard forms of therapy (including hydrodistension) or combination of therapies for PBS/IC.
* Participant will receive cystoscopy to be performed in the office at baseline visit before randomization if none has been conducted within the previous 24 weeks. Cystoscopy results must show no unevaluated lesions.
* Female participants with a cervix are required to have Pap smear exam within the past 12 months prior to enrollment with normal results reported.
* Participant (female) with child-bearing potential must agree to use two reliable/medically approved methods of birth control.

Exclusion Criteria:

* History of cancer or known pre-malignant conditions, including skin cancer.
* History of bladder calculus, tuberculous cystitis; neurologic disease affecting bladder function.
* Current immunocompromised condition, including current or chronic treatment with immunosuppressive agents, or known positive for HIV (positive antibody confirmed by Western Blot or IFA); active tuberculosis requiring on-going therapy; current systemic steroid treatment at any dose.
* Liver function test or creatinine results greater than 2x the upper limit of normal at home institution laboratory.
* Any baseline leukopenia (an absolute neutrophil count <1,500/µL), thrombocytopenia (a platelet count less than 150,000/microL), or anemia - HGB < 12 or < 11 g/dLin men and in women respectively.
* Is seropositive for Hepatitis B surface antigen; or is seropositive for Hepatitis B surface antibody (if not previously vaccinated); is seropositive for Hepatitis C antibody or HIV antigen or antibody.
* Allergy or hypersensitivity to study medication.
* Unable to void spontaneously.
* Active urethral or ureteral calculi, urethral diverticulum.
* Any severe debilitating or urgent concurrent medical condition.
* Previous cytoxan/cyclophosphamide treatment, pelvic radiation therapy; augmentation cystoplasty, cystectomy, or cystolysis; neurectomy.
* Participants with history of treatment for genital tract dysplasia or genital warts or genital herpes.
* Patients with active or a history of peptic ulcer disease, inflammatory bowel disease or gastrointestinal bleeding.
* Patients with hypertension not adequately controlled with medication.
* Patient currently taking H2 blockers or proton pump inhibitors.
* Patients who cannot tolerate or refuse an office cystoscopy.

Exclusion criteria for men only:

* Currently being treated for chronic bacterial prostatitis, as documented by a positive urine culture or prior history of recurrent bacterial urinary infections.
* Unevaluated suspicious prostate exam.

Exclusion criteria for women only:

* Lactation, pregnancy, or refusal of two types of (medically approved/reliable) birth control in women of child-bearing potential.
* Pain, frequency, urgency symptoms present only during menses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2007-03; Primary Completion 2008-02 (Actual); Study Completion 2008-04 (Estimated)

PRIMARY OUTCOMES:
To compare CellCept 2 grams daily to placebo for effects on overall IC symptoms and well being in patients with refractory PBS/IC. | 12 Weeks
To assess the safety profile of CellCept in the treatment of refractory PBS/IC. | 12 Weeks

SECONDARY OUTCOMES:
To investigate the association between clinical subgroups, characterized by differences in baseline characteristics (such as presence of ulcers, duration of symptoms, significant co-morbid diseases, serological abnormalities), and efficacy of CellCept. | 12 Weeks
To assess the patterns of patient expectations, associations with symptom severity, and the potential impact of patient expectations on response to treatment. | 12 Weeks
To assess patterns of treatment goals and goal achievement in this study population, as well as baseline characteristics and factors related to goal selection and achievement. | 12 Weeks
To assess impact of study medication on pain medication use. | 12 Weeks
To assess the frequency and mechanism of un-blinding on study results and assess how the patient's perception of which treatment they received changes over time and influences ultimate outcome. | 12 Weeks
To assess the rate of detectable immune disorders in patients with PBS/IC refractory to standard treatment using CellCept. | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Kusek, PhD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); LeRoy Nyberg, MD, PhD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); Richard Landis, PhD, Principal Investigator — University of Pennsylnania; David Burks, MD, Study Chair — Henry Ford Hospital; Harris Foster, MD, Principal Investigator — Yale University
Locations (11):
- United States (10):
  - Univeristy of California San Diego, San Diego, California
  - Stanford University Medical center, Stanford, California
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Maryland, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - University of Rochester, Rochester, New York
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - University of Washington, Seattle, Washington
- Queen's University, Kingston, Ontario, Canada

REFERENCES:
- See also: Interstitial Cystitis Association — http://www.ichelp.org/